CLINICAL TRIAL: NCT01125514
Title: A Single-blind, Multiple Dose, Placebo-controlled, Double Dummy Study to Investigate the Pharmacodynamic and Pharmacokinetic Interaction Between Aliskiren and Furosemide in Patients With Heart Failure
Brief Title: A Study to Investigate the Pharmacodynamic and Pharmacokinetic Interaction Between Aliskiren and Furosemide in Patients With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CSPP100A2255
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
Keywords: Heart failure,; aliskiren,; furosemide,; diuretic efficacy,; interaction
MeSH Terms: conditions — Heart Failure | interventions — aliskiren; Furosemide

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Furosemide 60 mg (Experimental): Treatment period 1 (Day 1 to Day 7): All eligible patients received 60 mg furosemide, 150 mg placebo of aliskiren, and 300 mg placebo aliskiren once daily.
  Interventions: Drug: Furosemide 60 mg; Drug: Placebo for Aliskiren
- Furosemide 60 mg + Aliskiren 150 mg (Experimental): Treatment Period 2 (Day 8 to day 17): Patients received 60 mg furosemide, 150 mg aliskiren and 300 mg placebo once daily.
  Interventions: Drug: Aliskiren 150 mg; Drug: Furosemide 60 mg; Drug: Placebo for Aliskiren
- Furosemide 60 mg + Aliskiren 300 mg (Experimental): Treatment Period 3 (Day 18 to day 27): Patients received 60 mg furosemide, 300 mg aliskiren and 150 mg placebo of aliskiren once daily.
  Interventions: Drug: Furosemide 60 mg; Drug: Placebo for Aliskiren; Drug: Aliskiren 300 mg

INTERVENTIONS:
Drug: Aliskiren 150 mg — Aliskiren 150 mg tablet
  Arms: Furosemide 60 mg + Aliskiren 150 mg
Drug: Furosemide 60 mg — Furosemide 60 mg commercially-available tablets
Drug: Placebo for Aliskiren — Matching placebo for aliskiren 150 mg and 300 mg
Drug: Aliskiren 300 mg — Aliskiren 300 mg tablet
  Arms: Furosemide 60 mg + Aliskiren 300 mg

SUMMARY:
This study assessed the interaction between single and multiple doses of aliskiren (150 mg and 300 mg) and furosemide (60 mg) in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Systolic or diastolic heart failure, diagnosed with either NYHA functional class II to III at least 3 months prior to screening and on stable medication for at least 12 weeks.
* Patients must have met either of the criteria at screening:
* Documented left ventricular ejection fraction (LVEF) greater than 20% but lower than 40% OR
* Patients with a documented LVEF greater than 40% and with a history of NT-pro-BNP> 400pg/mL (or BNP > 100pg/mL) within 12 months of screening.

Exclusion Criteria:

* Treatment with Angiotensin Receptor Blockers (ARBs), aldosterone receptor antagonists and diuretics (other than furosemide) within 3 weeks of first dose and during the study. Beta blockers were permitted provided the dose was stable for at least 3 weeks before the first dose and remains so throughout the study.
* Hypertrophic cardiomyopathy (HCMP).
* If a subject is currently treated with furosemide, the dose must be stable for at least 3 weeks before the first dose and the dose must not exceed 60 mg daily
* Stable heart failure requiring treatment with both an ACE inhibitor and an ARB or Current acute decompensated heart failure.
* Mean sitting systolic blood pressure ≥160 mmHg and/or mean sitting diastolic blood pressure ≥ 100mmHg and/or secondary forms of hypertension.
* Persistent sitting systolic blood pressure <90 mmHg.
* History of angioedema.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Vilnius, Lithuania

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide (Fu) /Fu+Aliskiren(Alis)150mg/fu+Alis 300mg: Treatment period 1 (Day 1 to Day 7): All eligible patients received 60 mg furosemide, 150 mg placebo of aliskiren, and 300 mg placebo aliskiren once daily.
  Treatment Period 2 (Day 8 to day 17): Patients received 60 mg furosemide, 150 mg aliskiren and 300 mg placebo once daily.
  Treatment Period 3 (Day 18 to day 27): Patients received 60 mg furosemide, 300 mg aliskiren and 150 mg placebo of aliskiren once daily.
  Day 28, no study treatment.
Period: Treatment Period 1 (Day 1 - Day 7)
Arm/Group | Furosemide (Fu) /Fu+Aliskiren(Alis)150mg/fu+Alis 300mg
Started | 37 (Randomized and safety population)
Completed | 35
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Administrative problems | 1
Period: Treatment Period 2 (Day 8 - Day 17)
Arm/Group | Furosemide (Fu) /Fu+Aliskiren(Alis)150mg/fu+Alis 300mg
Started | 35
Pharmacokinetic (PK) Analysis Set | 33
Pharmacodynamics (PD) Analysis Set | 33
Completed | 32
Not Completed | 3
Not completed — Adverse Event | 3
Period: Treatment Period2(Day9-Day27) and Day 28
Arm/Group | Furosemide (Fu) /Fu+Aliskiren(Alis)150mg/fu+Alis 300mg
Started | 32
Completed | 28
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Protocol Deviation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Furosemide (Fu) /Fu+Aliskiren(Alis)150mg/fu+Alis 300mg
Number analyzed (Participants) | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Diuretic Efficacy Index 1 for Sodium Excretion
Description: Efficacy of furosemide for sodium excretion (efficacy index 1) was defined by dividing urinary sodium excretion by the urinary excretion of furosemide. Diuretic index 1 for sodium was calculated for the for the total 0 to 4 hour urine collection.
Time Frame: 0 to 4 hours
Population: All patients who received at least one dose of study drug and had evaluable pharmacodynamic (PD) data with no major protocol deviation in at least one period were included in the PD analysis set.
Measure: Mean (Standard Deviation); unit: mmol/mg
Groups:
- Furosemide 60 mg + Aliskiren Placebo: Patient received 60 mg furosemide at steady state + placebo to aliskiren from day 1 to day 7.
- Furosemide 60 mg+ Single Dose Aliskiren 150mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 150mg on day 8.
- Furosemide 60 mg + Multiple Dose Aliskiren 150mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 150mg ( day 9 - day 17).
- Furosemide 60 mg + Multiple Dose Aliskiren 300mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 300mg ( day 18 - day 27).
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg+ Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 32 | 31 | 28
mmol/mg | 10.185 (4.4568) | 12.122 (6.2867) | 13.453 (8.3524) | 12.858 (6.1040)

2. Primary Outcome: Diuretic Efficacy Index 1 for Sodium Excretion
Description: Efficacy of furosemide for sodium excretion (efficacy index 1) was defined by dividing urinary sodium excretion by the urinary excretion of furosemide. Diuretic index 1 for sodium was calculated for the for the total 0 to 24 hour urine collection.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/mg
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg+ Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 31 | 31 | 30 | 28
mmol/mg | 10.775 (5.2486) | 13.264 (6.3535) | 13.364 (6.1511) | 14.747 (6.3531)

3. Secondary Outcome: Plasma Pharmacokinetics (PK) of Furosemide: Area Under the Plasma Concentration-time Curve (AUC)
Description: Pharmacokinetic (PK) parameters were determined from the plasma concentration time profile of furosemide using a non-compartmental method:
  AUCtau: Area under the plasma concentration-time curve from time zero to the end of the dosing interval
  AUC (0-24): Area under the plasma concentration-time curve from time zero to 24 hours
  AUClast: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. AUClast was calculated as the sum of linear trapezoids using non-compartmental analysis.
  AUCinf: Area under the plasma concentration-time curve from time zero to infinity. AUCinf was calculated by adding AUClast and the value obtained from dividing the last measurable plasma concentration by λz, where λz was determined from automated linear regression of the last three time points with non-zero concentrations in the terminal phase of the log-transformed concentration-time profile
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: All patients who received at least one dose of study drug and had evaluable Pharmacokinetic (PK) data with no major protocol deviation in at least one period were included in the PK analysis set.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Furosemide 60 mg + Single Dose Aliskiren 150mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 150mg on day 8.
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
h*ng/mL
  AUCtau | 5217 (1996.7) | 4255 (1390.6) | 4638 (1532.9) | 4218 (1469.3)
  AUC | 5217 (1996.7) | 4255 (1390.6) | 4638 (1532.9) | 4218 (1469.3)
  AUClast | 5154 (1999.2) | 4207 (1387.5) | 4535 (1531.6) | 4130 (1525.4)
  AUCinf | 5420 (2005.2) | 4559 (1387.4) | 4783 (1611.7) | 4381 (1578.3)

4. Secondary Outcome: Plasma Pharmacokinetics (PK) of Furosemide: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax, ss)
Description: Cmax,ss was directly determined from the raw plasma concentration-time data.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
ng/mL | 1702 (708.66) | 1326 (518.15) | 1317 (542.73) | 1180 (404.92)

5. Secondary Outcome: Plasma Pharmacokinetics (PK) of Furosemide: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Tmax was directly determined from the raw plasma concentration-time data.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: All patients who received at least one dose of study drug and had evaluable PK data with no major protocol deviation in at least one period were included in the PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
Hours | 1.500 [1.00 to 3.00] | 1.500 [0.500 to 3.00] | 1.500 [1.00 to 4.00] | 2.00 [0.500 to 3.00]

6. Secondary Outcome: Plasma Pharmacokinetics (PK) of Furosemide: Average Steady State Plasma Concentration During Multiple Dosing (Cav,ss)
Description: The average steady-state drug concentration in the plasma, blood, serum, or other body fluids during multiple dosing [amount x volume-1]. This was estimated as AUCτ/τ
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: All subjects with evaluable pharmacokinetic parameter data with no exclusion flags and no major protocol deviations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
ng/mL | 217.4 (83.196) | 177.3 (57.942) | 193.2 (63.872) | 175.8 (61.219)

7. Secondary Outcome: Plasma Pharmacokinetics (PK) of Furosemide: Lowest Plasma Concentration Observed During a Dosing Interval at Steady State (Cmin, ss)
Description: The minimum observed steady-state drug concentration in the plasma, blood, serum, or other body fluids at the end of the dosing interval during multiple dosing [amount x volume-1]
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Furosemide 60 mg+ Multiple Dose Aliskiren 150mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 150mg ( day 9 - day 17).
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg+ Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
ng/mL | 20.42 (25.558) | 20.03 (23.780) | 19.80 (29.258) | 16.70 (20.868)

8. Secondary Outcome: Urine Pharmacokinetics (PK) of Furosemide: Amount of Drug Excreted Into the Urine From Time Zero to 24 Hours After Administration (Ae0-24)
Description: The area under the plasma (or serum or blood) concentration-time curve from time zero to 24 h [mass × time × volume-1]
Time Frame: 0 to 4, 4 to 8, 8 to 12 and 12 to 24 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Furosemide 60 mg+ Multiple Dose Aliskiren 300mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 300mg ( day 18 - day 27).
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg+ Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 31 | 31 | 30 | 28
mg | 18.61 (5.9012) | 15.08 (3.9613) | 14.98 (4.5264) | 13.63 (4.5134)

9. Secondary Outcome: Urine Pharmacokinetics (PK) of Furosemide: Renal Clearance (CLR)
Description: The renal clearance of drug [volume x time-1]
Time Frame: 0 to 4, 4 to 8, 8 to 12 and 12 to 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 31 | 31 | 30 | 28
L/h | 3.808 (1.3567) | 3.841 (1.4321) | 3.519 (1.3592) | 3.561 (1.4458)

10. Secondary Outcome: Creatinine Clearance
Description: Creatinine clearance= (Urine creatinine/Serum creatinine) x (Urine volume/(24*60)).
Time Frame: 0 to 4, 4 to 8, 8 to 12 and 12 to 24 hours post dose
Population: All patients who received at least one dose of study drug and had evaluable PD data with no major protocol deviation in at least one period were included in the PD analysis set.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 32 | 32 | 29 | 28
mL/min | 104.745 (38.2884) | 109.657 (30.0667) | 103.841 (28.2845) | 105.304 (25.4076)

11. Secondary Outcome: Urine Sodium and Potassium Excretion Per Treatment at 4 Hours Postdose
Description: Urine was collected 4 hours postdose in all treatment groups for sodium and potassium analysis. Each patient was required to void their bladder before drug administration and at the end 4 hours.
Time Frame: 4 hours postdose
Population: All patients who received at least one dose of study drug and had evaluable pharmacodynamics (PD)data with no major protocol deviation in at least one period were included in the PD analysis set.
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 32 | 31 | 28
mmol
  Sodium excretion | 113.992 (47.5976) | 104.031 (49.5036) | 98.691 (55.0495) | 93.341 (43.9419)
  Potassium excretion | 24.555 (11.9749) | 19.403 (10.5975) | 23.046 (8.6829) | 21.037 (7.9355)

12. Secondary Outcome: Urine Sodium and Potassium Excretion Per Treatment at 8 Hours Postdose
Description: Urine was collected 8 hours postdose in all treatment groups for sodium and potassium analysis. Each patient was required to void their bladder before drug administration and at the end 8 hours.
Time Frame: 8 hours postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 31 | 31 | 28
mmol
  Sodium excretion | 129.990 (49.2835) | 123.835 (56.2734) | 125.677 (58.6125) | 119.776 (59.0523)
  Potassium excretion | 33.474 (12.2417) | 28.068 (12.5292) | 36.120 (14.4509) | 32.498 (9.6174)

13. Secondary Outcome: Urine Sodium and Potassium Excretion Per Treatment at 12 Hours Postdose
Description: Urine was collected 12 hours postdose in all treatment groups for sodium and potassium analysis. Each patient was required to void their bladder before drug administration and at the end 12 hours.
Time Frame: 12 hours postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 32 | 32 | 31 | 27
mmol
  Sodium excretion | 151.254 (57.6190) | 142.476 (59.1617) | 144.839 (63.6708) | 140.887 (68.4341)
  Potassium excretion | 45.013 (17.3416) | 37.827 (16.0087) | 46.770 (17.4395) | 44.137 (11.0631)

14. Secondary Outcome: Urine Sodium and Potassium Excretion Per Treatment at 24 Hours Postdose
Description: Urine was collected 24 hours postdose in all treatment groups for sodium and potassium analysis. Each patient was required to void their bladder before drug administration and at the end 24 hours.
Time Frame: 24 hours postdose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 31 | 31 | 30 | 28
mmol
  Sodium excretion | 185.426 (69.9537) | 187.256 (69.1028) | 188.886 (73.8708) | 192.176 (76.0983)
  Potassium excretion | 57.323 (20.0607) | 53.107 (21.3416) | 62.715 (20.4014) | 61.012 (13.6072)

15. Secondary Outcome: Mean Sitting Systolic Blood Pressure (msSBP)and Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting blood pressure was measured three times at 1 to 2-minute intervals. The mean of the three sitting blood pressure measurements was used as the average of the sitting office blood pressure. The msSBP and msDBP data were analyzed using a mixed effect model with fixed effects from treatment and treatment*time; random effect from patients and predose as covariate.
Time Frame: 0.5 hour pre-dose, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose.
Population: Safety analysis set include subjects that received study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Furosemide go mg + Multiple Dose Aliskiren 300mg: Patient received 60 mg furosemide at steady state + single dose aliskiren 300mg ( day 18 - day 27).
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide go mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 37 | 35 | 32
mmHg
  0.5 predose (msSBP) | 118.26 (1.62) | 117.09 (1.70) | 116.63 (1.80)
  0.5 hour predose (msDBP) | 71.70 (0.98) | 71.41 (1.04) | 71.39 (1.10)
  0.5 hour Postdose (msSBP) | 114.78 (1.64) | 113.19 (1.70) | 114.31 (1.80)
  0.5 hour Postdose (msDBP) | 70.94 (1.00) | 69.04 (1.04) | 69.86 (1.10)
  1 hour Postdose (msSBP) | 115.15 (1.64) | 112.22 (1.70) | 112.16 (1.80)
  1 hour Postdose (msDBP) | 71.22 (1.00) | 69.04 (1.04) | 68.96 (1.10)
  2 hour Postdose (msSBP) | 113.61 (1.64) | 109.22 (1.70) | 109.63 (1.80)
  2 hour Postdose (msDBP) | 68.39 (1.10) | 67.50 (1.04) | 68.39 (1.10)
  4 hour Postdose (msSBP) | 106.50 (1.64) | 101.84 (1.70) | 101.06 (1.80)
  4 hour Postdose (msDBP) | 63.85 (1.00) | 62.32 (1.04) | 59.07 (1.10)
  8 hour Postdose (msSBP) | 110.75 (1.66) | 112.09 (1.70) | 109.95 (1.80)
  8 hour Postdose (msDBP) | 66.33 (1.01) | 66.94 (1.04) | 66.46 (1.10)
  12 hour Postdose (msSBP) | 116.99 (1.66) | 116.90 (1.70) | 115.16 (1.80)
  12 hour Postdose (msdBP) | 67.86 (1.01) | 68.79 (1.04) | 68.50 (1.10)
  24 hour Postdose (msSBP) | 115.49 (1.66) | 116.69 (1.72) | 118.41 (1.80)
  24 hour Postdose (msDBP) | 71.24 (1.01) | 71.66 (1.05) | 72.32 (1.10)

16. Primary Outcome: Diuretic Efficacy Index 2 for Water Excretion
Description: Efficacy of furosemide for water excretion (efficacy index 2) was defined by dividing urine volume by the urinary excretion of furosemide.Diuretic index 2 for water was calculated for the 0 to 4 hour fraction urine collection.
Time Frame: 0 to 4 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mL/mg
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 33 | 32 | 31 | 28
mL/mg | 90.402 (34.7866) | 109.773 (50.2433) | 119.239 (63.3655) | 122.157 (58.8815)

17. Primary Outcome: Diuretic Efficacy Index 2 for Water Excretion
Description: Efficacy of furosemide for water excretion (efficacy index 2) was defined by dividing urine volume by the urinary excretion of furosemide.Diuretic index 2 for water was calculated for the 0 to 4 hour fraction and for the total 0 to 24 hour urine collection.
Time Frame: 0 to 24 hours
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mL/mg
Arm/Group | Furosemide 60 mg + Aliskiren Placebo | Furosemide 60 mg + Single Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 150mg | Furosemide 60 mg + Multiple Dose Aliskiren 300mg
Number analyzed (Participants) | 31 | 32 | 30 | 28
mL/mg | 119.439 (46.2607) | 151.859 (53.6734) | 154.116 (40.5598) | 175.112 (59.4236)

ADVERSE EVENTS:
Groups:
- 60 mg Furosemide + 150 mg Placebo + 300 mg Placebo: 60 mg furosemide + 150 mg placebo + 300 mg placebo
- 60 mg Furosemide + 150 mg Aliskiren + 300 mg Placebo: 60 mg furosemide + 150 mg aliskiren + 300 mg placebo
- 60 mg Furosemide + 300 mg Aliskiren + 150 mg Placebo: 60 mg furosemide + 300 mg aliskiren + 150 mg placebo
Arm/Group | 60 mg Furosemide + 150 mg Placebo + 300 mg Placebo | 60 mg Furosemide + 150 mg Aliskiren + 300 mg Placebo | 60 mg Furosemide + 300 mg Aliskiren + 150 mg Placebo
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg Furosemide + 150 mg Placebo + 300 mg Placebo (N=37) | 60 mg Furosemide + 150 mg Aliskiren + 300 mg Placebo (N=33) | 60 mg Furosemide + 300 mg Aliskiren + 150 mg Placebo (N=31)
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.